CLINICAL TRIAL: NCT03337386
Title: Reliability of Subclavian Vein Versus Inferior Vena Cava Collapsibility Indices for Preload Assessment.
Brief Title: Subclavian Versus Inferior Vena Cava Collapsibility Indices.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Alaa Mazy Mazy, Associate professor of anesthesia and surgical intensive care, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS/17.05.137
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Central Venous Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inferior Vena Cava Collapsibility (Experimental): inferior vena cava diameters is obtained in the supine position with a convex probe .The probe is placed in the subxiphoid region or the right anterior midaxillary plane.The sagittal section of IVC is imaged. M-mode probe is used to identify the measurement of minimum and maximum venous dimensions over the respiratory cycle using the 3.5-5 MHz phased array probe. To standardize the measurements, measuring of the IVC diameter is performed at 2 cm caudal of the junction point of the right atrium and IVC. The difference between the maximum (D max) and minimum (D min)diameters of the target vein is normalized according to the standard formula to yield the collapsibility index (CI).
  Interventions: Diagnostic Test: inferior vena cava collapsibility
- Subclavian Vein Collapsibility (Experimental): Right SCV diameters is checked in the supine position using a high frequency linear array probe (6-13 MHz) and M-mode. To standardize the measurements, the probe is placed beneath the proximal part of the middle part of the clavicle perpendicular to long-axis of the SCV to obtain the best cross-sectional view of the vien. After the target vein is localized , the dynamic diameter change is recorded using M-mode to identify and measure the minimum and maximum venous diameters.To calculate SCV collapsibility index, the standard formula is used.
  Interventions: Diagnostic Test: subclavian vein collapsibility
- central venous pressure (Active Comparator): ultrasound guided 7.5-F central venous catheter is introduced via right internal jugular vein under local analgesia with 2% lidocaine for measuring the CVP.
  Interventions: Diagnostic Test: central venous pressure

INTERVENTIONS:
Diagnostic Test: inferior vena cava collapsibility — inferior vena cava diameters is obtained in the supine position with a convex probe .The probe is placed in the subxiphoid region or the right anterior midaxillary plane.The sagittal section of IVC is imaged. M-mode probe is used to identify the measurement of minimum and maximum venous dimensions over the respiratory cycle using the 3.5-5 MHz phased array probe. To standardize the measurements, measuring of the IVC diameter is performed at 2 cm caudal of the junction point of the right atrium and IVC. The difference between the maximum (D max) and minimum (D min)diameters of the target vein is normalized according to the standard formula to yield the collapsibility index (CI).
  Arms: Inferior Vena Cava Collapsibility
Diagnostic Test: subclavian vein collapsibility — Right SCV diameters is checked in the supine position using a high frequency linear array probe (6-13 MHz) and M-mode. To standardize the measurements, the probe is placed beneath the proximal part of the middle part of the clavicle perpendicular to long-axis of the SCV to obtain the best cross-sectional view of the vien. After the target vein is localized , the dynamic diameter change is recorded using M-mode to identify and measure the minimum and maximum venous diameters.To calculate SCV collapsibility index, the standard formula is used.
  Arms: Subclavian Vein Collapsibility
Diagnostic Test: central venous pressure — ultrasound guided 7.5-F central venous catheter is introduced via right internal jugular vein under local analgesia with 2% lidocaine for measuring the CVP.
  Arms: central venous pressure

SUMMARY:
Traditional methods for intravascular volume status assessment include physical examination, raised leg test, central venous pressure (CVP) and pulmonary artery catheters occlusion pressure (PAWP). Central venous pressure and pulmonary artery occlusion pressure are invasive and associated with significant complications. More recently, a number of less invasive techniques have been introduced, but they lack standardization and reliability. Ultrasonically, inferior vena cava collapsibility can detect hypovolemia non-invasively.

DETAILED DESCRIPTION:
The aim of this study is that measurement of subclavian vein collapsibility index(SCV-CI) could be potential adjunct to IVC-CI where the IVC visualization is impaired or not possible .

-Finding a non-invasive reliable accurate method for evaluation of intravascular volume and response to volume resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* 1. American society of anaesthesiologists physical status grade I and grade II .

  2. Elective laparotomy. 3. Supine position

Exclusion Criteria:

1. Patient refusal .
2. Portal hypertension .
3. Severe peripheral vascular diseases.
4. Obstructive lung diseases .
5. Right sided heart failure , arrhythmia and valvular heart heart diseases .
6. Body mass index >35 kg/m2

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-12 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
inferior vena cava collapsibility index changes | intraoperative changes:1st basal before induction of anesthesia, 2nd before start of surgery, 3rd after10 ml/kg ringers preload, 4th 5 minutes before extubation.
  ultrasound M mode maximum minus minimum over maximum then multiply by 100

SECONDARY OUTCOMES:
subclavian vein collapsibility index changes | intraoperative changes:1st basal before induction of anesthesia, 2nd before start of surgery, 3rd after 10 ml/kg ringers preload, 4th 5 minutes before extubation.
  ultrasound M mode maximum minus minimum over the maximum then multiply by 100
central venous pressure changes | intraoperative changes:1st basal before induction of anesthesia, 2nd before start of surgery, 3rd after 10 ml/kg ringers preload, 4th 5 minutes before extubation.
  centimeter water
heart rate changes | intraoperative changes:1st basal before induction of anesthesia, 2nd before start of surgery, 3rd after 10 ml/kg ringers preload, 4th 5 minutes before extubation.
  beat per minute
mean blood pressure changes | intraoperative changes:1st basal before induction of anesthesia, 2nd before start of surgery, 3rd after 10 ml/kg ringers preload, 4th 5 minutes before extubation.
  millimeter mercury
fluid administration | Intraoperative
  milliliter
blood loss | intraoperative
  milliliter
urine output | intraoperative
  milliliter

CONTACTS AND LOCATIONS:
Locations (1):
- Oncolgy Center, Mansoura University,, Al Mansurah, DK, Egypt